CLINICAL TRIAL: NCT04365465
Title: BRIDGE Device: Percutaneous Auricular Nerve Field Stimulation as Alternative Post-Cesarean Delivery Analgesia
Brief Title: BRIDGE Percutaneous Nerve Stimulation for Cesarean Delivery Pain Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Grace Lim, MD, MS (Other)
Collaborators: University of Pittsburgh (Other)
Responsible Party: Sponsor-Investigator, Grace Lim, MD, MS, Assistant Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STUDY19110257; UL1TR001857 (NIH)
Record Dates: First submitted 2020-04-21; First posted 2020-04-28 (Actual); Results first posted 2023-01-18 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2022-12

CONDITIONS: Opioid-use Disorder; Pain, Postoperative
MeSH Terms: conditions — Opioid-Related Disorders; Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: This study is a randomized control trial with the following arms: 1) active device; 2) placebo device; 3) non-intervention (active control).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Among participants who receive a device, both the participant and care providers/investigators will be blinded to whether the device is active or placebo. There is no blinding among participants who do not receive a device.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Active device (Experimental): Participants in this arm will receive an active NSS-Bridge device placed immediately following their cesarean section.
  Interventions: Device: NSS-2 Bridge
- Placebo device (Sham Comparator): Participants in this arm will receive an inactive (sham) NSS-Bridge device placed immediately following their cesarean section.
  Interventions: Device: Inactive NSS-2 Bridge
- Active Control (Active Comparator): Participants in this arm will receive no device, only the standard postpartum pain control.
  Interventions: Other: Active control

INTERVENTIONS:
Device: NSS-2 Bridge — The NSS-2 BRIDGE (Appendix 1) is a battery operated and disposable percutaneous auricular nerve field stimulator (Innovative Health Solutions, Versailles, IN, USA), that was recently cleared by the FDA and assigned a Class II Risk Designation; a class which includes surgical drapes, pumps and power wheelchairs.
  Arms: Active device
Device: Inactive NSS-2 Bridge — This is a sham device which is identical to the active NSS-2 Bridge, but will not provide percutaneous auricular nerve field stimulation when applied.
  Arms: Placebo device
Other: Active control — Active control will include standard of care pain management during the postoperative period. Participants in this intervention arm will not receive or wear a device.
  Arms: Active Control

SUMMARY:
This is a randomized, placebo controlled and natural-history controlled trial to investigate the effectiveness of NSS-2 BRIDGE® for postpartum women with AND without opioid use disorder (OUD). The purpose of this pilot investigation is to establish feasibility/acceptability of the trial design.

DETAILED DESCRIPTION:
This study is a randomized control trial with the following arms: 1) active device; 2) placebo device; 3) non-intervention (active control). The devices will be placed while women are still feeling pain relief from labor epidural analgesia (after delivering vaginally) or from spinal or epidural anesthesia (after delivering by cesarean). By applying the devices while women are still relatively pain-free, a preventative/pre-emptive approach to pain management in women at risk for severe postpartum pain is taken. The study will enroll women with and without OUD and follow them for five days postpartum.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant
* Third trimester
* Cesarean delivery under neuraxial anesthesia
* Healthy, clean skin
* 18 years or older

Exclusion Criteria:

* Not fluent in English (surveys are validated in English language), unable to participate in informed consent discussions, or unable to give informed consent for any reason
* Unable to participate fully in all study procedures for any reason
* Cesarean delivery under general anesthesia
* History of hemophilia
* Pacemakers or implantable electronic devices
* History of psoriasis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-08-17 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Grace Lim, MD, MS, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Magee Womens Hospital, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active Device | Placebo Device | Active Control
Started | 20 | 20 | 20
Completed | 20 | 20 | 20
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Device | Placebo Device | Active Control | Total
Number analyzed (Participants) | 20 | 20 | 20 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 20 | 20 | 20 | 60
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.7 (5.5) | 32.1 (4.7) | 31.4 (5.8) | 32.07 (0.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 20 | 20 | 60
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1 | 2
  Not Hispanic or Latino | 20 | 18 | 17 | 55
  Unknown or Not Reported | 0 | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 2 | 5
  White | 18 | 17 | 17 | 52
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 20 | 60
Education Level [Count of Participants; unit: Participants]
  High school graduate, diploma, or equivalent | 4 | 1 | 1 | 6
  Trade, technical, vocational training | 1 | 3 | 3 | 7
  Some college credit, no degree | 3 | 3 | 3 | 9
  Associate degree | 3 | 1 | 1 | 5
  Bachelor's degree | 3 | 2 | 2 | 7
  Master's degree | 1 | 5 | 4 | 10
  Doctorate degree | 0 | 0 | 0 | 0
  Unknown or Not Reported | 5 | 5 | 6 | 16
Income Level [Count of Participants; unit: Participants]
  Less than $10,000 | 1 | 2 | 2 | 5
  $10,000 to $19,999 | 2 | 0 | 1 | 3
  $20,000 to $29,999 | 1 | 2 | 1 | 4
  $30,000 to $39,999 | 1 | 0 | 0 | 1
  $40,000 to $49,999 | 1 | 1 | 1 | 3
  $50,000 to $59,999 | 1 | 0 | 0 | 1
  $60,000 to $69,999 | 2 | 2 | 0 | 4
  $70,000 to $79,999 | 0 | 2 | 4 | 6
  $80,000 to $89,999 | 2 | 3 | 1 | 6
  $90,000 to $99,999 | 1 | 4 | 1 | 6
  $100,000 to $149,999 | 6 | 2 | 3 | 11
  $150,000 or more | 2 | 2 | 5 | 9
  Unknown or Not Reported | 0 | 0 | 1 | 1
Body Mass Index [Median (Inter-Quartile Range); unit: kg/m^2] | 31.9 [21.88 to 44.4] | 29.7 [25.8 to 34.5] | 34.8 [24.2 to 51.9] | 31.9 [21.88 to 51.9]
Gravidity [Median (Inter-Quartile Range); unit: Number of pregnancies] | 2 [1 to 5] | 2.5 [1 to 8] | 2 [1 to 8] | 2 [1 to 8]
Parity [Mean (Inter-Quartile Range); unit: Number of offspring] | 1 [0 to 2] | 1 [0 to 3] | 1 [0 to 5] | 1 [0.68 to 1.16]
History of Anxiety/Depression [Count of Participants; unit: Participants] | 14 | 10 | 10 | 34
History of Mental Illness [Count of Participants; unit: Participants] | 4 | 3 | 1 | 8
Prior Cesareans [Median (Inter-Quartile Range); unit: Number of prior cesareans] | 1 [0 to 2] | 1 [0 to 3] | 1 [0 to 5] | 1 [0.58 to 1.06]
Opioid Use Disorder [Count of Participants; unit: Participants] | 0 | 0 | 1 | 1
Medication for Opioid Use Disorder [Count of Participants; unit: Participants] | 0 | 0 | 1 | 1
Substance Use Disorder [Count of Participants; unit: Participants] | 4 | 1 | 3 | 8

OUTCOME MEASURES:

1. Primary Outcome: Pain Scores With Movement
Description: Pain Score with movement will be measured by a score on a scale (0=no pain 10=most pain). The minimum value is 0 and the maximum value is 10. Higher scores mean a worse outcome.
Time Frame: post-operative day 3
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Active Device | Placebo Device | Active Control
Number analyzed (Participants) | 20 | 20 | 20
score on a scale | 4.57 (0.231) | 4.61 (0.234) | 4.19 (.229)

2. Secondary Outcome: PROMIS Pain Intensity Survey
Description: PROMIS Pain Intensity Survey is self-reported by participants and includes the options: "Had no pain", "Mild", "Moderate", "Severe", or "Very Severe". These responses range from 1 point (had no pain) to 5 points (very severe). This means the participant raw score can be between 3 points and 15 points.
Time Frame: Post-operative day 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Device | Placebo Device | Active Control
Number analyzed (Participants) | 20 | 20 | 20
score on a scale | 8.23 (2.04) | 7.9 (2.05) | 7.8 (1.79)

3. Secondary Outcome: PROMIS Pain Interference Survey
Description: PROMIS Pain Interference Survey is self-reported by participants and includes the options: "Not at all", "A little bit", "Somewhat", "Quite a bit", or "Very Much". These responses range from 1 point (not at all) to 5 points (very much). This means the participant raw score can be between 3 points and 15 points.
Time Frame: Post-operative day 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Device | Placebo Device | Active Control
Number analyzed (Participants) | 20 | 20 | 20
score on a scale | 9.47 (3.52) | 9.0 (3.42) | 9.0 (3.11)

4. Secondary Outcome: Opioid Consumption
Description: Total opioid consumption as abstracted from EMR during hospital stay. The number of participants using opioids by post-operative day 3 will be recorded by binary responses of 'yes' or 'no' via EMR data.
Time Frame: Post-operative day 3
Measure: Count of Participants; unit: Participants
Arm/Group | Active Device | Placebo Device | Active Control
Number analyzed (Participants) | 20 | 20 | 20
Participants
  Opioid-free | 8 | 4 | 6
  Used opioids | 12 | 16 | 14

5. Secondary Outcome: ObsQoR-11 Survey
Description: 11 item survey evaluation of postoperative symptoms and independence as self reported by participants. Scale for this tool is 0-10 with 0 being "very poor" and 10 being "excellent". Total score will be calculated for each participant. Minimum score = 0 and Maximum score = 110
Time Frame: Post-operative day 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Device | Placebo Device | Active Control
Number analyzed (Participants) | 20 | 20 | 20
score on a scale | 79.32 (20.85) | 76.9 (21.47) | 80.3 (17.9)

6. Secondary Outcome: Recovery Variables From Med Record: ICU Admission
Description: ICU admission as abstracted from EMR during hospital stay. This will be recorded with a binary response of 0. no or 1. yes if participant is admitted to the ICU in the first week post-op.
Time Frame: First week postoperatively
Measure: Count of Participants; unit: Participants
Arm/Group | Active Device | Placebo Device | Active Control
Number analyzed (Participants) | 20 | 20 | 20
Participants | 0 | 0 | 0

7. Secondary Outcome: Recovery Variables From Med Record: Readmission
Description: Readmission as abstracted from EMR during hospital stay.
Time Frame: First week postoperatively
Measure: Count of Participants; unit: Participants
Arm/Group | Active Device | Placebo Device | Active Control
Number analyzed (Participants) | 20 | 20 | 20
Participants | 0 | 0 | 0

8. Secondary Outcome: Recovery Variables From Med Record: Readmission Due to Pain Issues
Description: Readmission due to pain issues as abstracted from EMR during hospital stay.
Time Frame: First week postoperatively
Measure: Count of Participants; unit: Participants
Arm/Group | Active Device | Placebo Device | Active Control
Number analyzed (Participants) | 20 | 20 | 20
Participants | 0 | 0 | 0

9. Secondary Outcome: BPI8 Survey
Description: 1 item survey of percentage of relief experienced from pain management as self-reported by participants. Percentage options: 0, 10, 20, 30, 40, 50, 60, 70, 80, 90, 100. Participant will self-report on post-operative day 3. Percentages will be converted to a 0-10 scale. A score of 0 (minimum value) indicates better outcomes and a score of 10 (maximum value) indicates worse outcomes
Time Frame: Post-operative day 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Device | Placebo Device | Active Control
Number analyzed (Participants) | 20 | 20 | 20
score on a scale | 8.5 (1.77) | 8.3 (2.10) | 2.9 (2.37)

10. Secondary Outcome: BPI25 Survey
Description: 1 item survey of pain medication use frequency as self-reported by participants. Scored on a 1-5 scale, with 1 indicating better outcomes and 5 indicating worse outcomes.
Time Frame: Post-operative day 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Device | Placebo Device | Active Control
Number analyzed (Participants) | 20 | 20 | 20
score on a scale | 2.91 (0.41) | 2.93 (0.56) | 2.93 (0.56)

11. Secondary Outcome: Device Tolerability Survey
Description: Device tolerability will be recorded using a Visual Analogue Scale (VAS). This will be self-reported by participants. Response options: 0, 10, 20, 30, 40, 50, 60, 70, 80, 90, or 100. 0 = no pain at all and 100 = severe intolerable pain.
Time Frame: Post-Op Day 7
Measure: Mean (Standard Deviation); unit: VAS Score
Arm/Group | Active Device | Placebo Device
Number analyzed (Participants) | 20 | 20
VAS Score | 76.8 (22.1) | 80.1 (20.0)

ADVERSE EVENTS:
Time Frame: Active participation was from day of surgery to 1-week post-operative. During this time period, adverse events were monitored and recorded.
Arm/Group | Active Device | Placebo Device | Active Control
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-02-02): https://cdn.clinicaltrials.gov/large-docs/65/NCT04365465/Prot_SAP_004.pdf
  • Informed Consent Form (2021-02-24): https://cdn.clinicaltrials.gov/large-docs/65/NCT04365465/ICF_006.pdf